CLINICAL TRIAL: NCT00168883
Title: Randomized Phase II Study to Determine the Efficacy of a Three Weekly vs. Weekly Therapy With Paclitaxel Plus Carboplatin vs. Paclitaxel Plus Vinorelbine for Patients With Non Small Cell Lung Cancer According to UICC Stage IIIB and IV
Brief Title: Study for Patients With Non Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Bristol-Myers Squibb (Industry); Pierre Fabre Pharma GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Haema CBF NSCLC UK/AS 03
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2006-11-01 (Estimated); Status verified 2006-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC; curative non-treatable NSCLC UICC stage IIIB and IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Vinorelbine

INTERVENTIONS:
Drug: Carboplatin
Drug: Paclitaxel
Drug: Vinorelbine

SUMMARY:
This is a randomized study to assess the efficacy and safety of chemotherapy with platin compared to chemotherapy without platin.

DETAILED DESCRIPTION:
Randomized Phase II design, multicenter study, to assess the efficacy and safety of combined chemotherapy with Paclitaxel and Carboplatin versus a platinum free chemotherapy with Paclitaxel and Vinorelbine, within the combination therapies there are two different dosing intervals, which will be assessed as well (4 Arm study).

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy naive patients with histologically confirmed NSCLC stage III and IV

Exclusion Criteria:

* New York Heart Association (NYHA) III or IV
* Brain metastases
* Neurotoxicity Grade 2 or greater

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2002-10; Study Completion 2006-12

PRIMARY OUTCOMES:
Determination of response rate (stable disease [SD] or better)
Determination of safety of the combination and life quality

SECONDARY OUTCOMES:
Determination of remission rate
Determination of time to progression
Determination of 1-year survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Keilholz, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Hematology & Oncology Charité CBF Berlin, Berlin, State of Berlin, Germany